CLINICAL TRIAL: NCT01758991
Title: Therapeutic Impact of tDCS on Dysphagia in the Acute Phase of Stroke / Impact thérapeutique de la tDCS Sur la Dysphagie en Phase Aigue de l'Accident Vasculaire cérébral
Brief Title: Improving SWAllowing After Stroke With Transcranial Direct Current Stimulation
Acronym: iSWAT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: University Hospital of Mont-Godinne (Other)
Collaborators: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Pr Yves Vandermeeren, MD, PhD, Professor (MD, PhD), University Hospital of Mont-Godinne
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B039201111926
Record Dates: First submitted 2012-12-27; First posted 2013-01-01 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Acute Stroke; Dysphagia
MeSH Terms: conditions — Stroke; Deglutition Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: tDCS
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: randomisation by computer
Oversight: Data Monitoring Committee: No

ARMS (2):
- real tDCS (Active Comparator): patients will receive non-invasive and painless brain stimulation over the rain areas involved in swallowing.
  tDCS will be applied during swallowing therapy, during 20 minutes
  Interventions: Device: transcranial direct current stimulation (tDCS)
- sham tDCS (Placebo Comparator): this will be exactly as for "real tDCS" unless that the tDCS will be rapidly turned off, unbeknown from patients-therapist-examinator (double-blind trial)
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — tDCS is a safe and painless transcranial stimulation that modulates brain activity and could improve stroke recovery. Electrodes in soaked sponges are placed over specific brain regions and held with an elastic band. Direct current is then applied through the electrodes. The patients may feel nothing or a slight tingling under the electrodes.
  Other Names: Eldith PLUS tDCS, NeuroConn, Ilmenau, Germany

SUMMARY:
In the acute phase of stroke, dysphagia (difficulty/inability to swallow) is a common problem that can have serious consequences such as aspiration pneumonia, increased lenght of hospitalisation, and death. It would be interesting to enhance the therapeutic effect of swallowing retraining by means on non-invasive brain stimulation such as transcranial direct current stimulation (tDCS).

Hypothesis: during the acute phase of stroke, applying tDCS over the brain during the revalidation and/or supervised feeding improves dysphagia significantly when compared to sham tDCS.

DETAILED DESCRIPTION:
tDCS will be used in a double-blind, randomized control trial in acute stroke patients suffering from dysphagia.

After informed consent and recruitment, patients will be randomly (computer method) allocated to real or sham tDCS, that will be applied during swallowing exercices/therapy or supervised feeding.

Baseline and follow-up outcomes about dysphagia will be collected.

ELIGIBILITY:
Inclusion Criteria:

- acute stroke (ischemic / hemorrhagic) with dysphagia

Exclusion Criteria:

* major swallowing impairment before the stroke
* troubles of comprehension impairing communication
* major cognitive dysfunction, neuro-degenerative disease, or major psychiatric condition (e.g. depression, Alzheimer's disease, …)
* very unstable health issue (e.g. severe cardiac dyscfct, end-stage renal failure, unstable diabetes, …)
* intracranial metal and/or devices excluding tDCS application
* chronic intake of major drugs modifying brain activity (e.g. AEDs, antipsychotics)
* regular use of alcohol or recreative drugs
* epilepsy
* pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2023-05-08 (Actual); Study Completion 2023-05-08 (Actual)

PRIMARY OUTCOMES:
VideoFluoroscopy (VFSS) | baseline, end of acute stroke phase, follow up (3, 6, 12 months)
  The patients will be asked to swallow radiocontrast agent liquid during RX (radiography) video-recording. The speed of swallowing, whether there is aspiration or stasis will be quantified off-line on videotape
Fiberoptic Endoscopic Evaluation of Swallowing (FEES) | baseline, end of acute stroke phase, follow up (3, 6, 12 months)
  A laryngoscope (attached to a camera and a color monitor) will be passed through the nostril.
  The patients will be asked to swallow small quantities of liquids and foods, and the quality of swallowing will be assessed off-line (videotaped examination).
  The base of the tongue, pharynx and larynx will be viewed.

SECONDARY OUTCOMES:
NIH Stroke Scale | baseline, end of acute stroke phase, follow up (3, 6, 12 months)
  The NIS Stroke Scale is a clinical scale developped to score the severity of acute stroke. Patients will be asked to make some movements, vision will be tested, whether there are difficult to speak and so on.
clinical record | baseline, end of acute stroke phase, follow up (3, 6, 12 months)
  the records of the acute stroke patients will be used to search for relevant clinical events.
quality-of-life (QOL) questionnaire designed for dysphagia (SWAL-QOL) | baseline, end of acute stroke phase, follow up (3, 6, 12 months)
  A quality-of-life (QOL) questionnaire specifically designed for patients with oropharyngeal dysphagia (SWAL-QOL) will be used, questions will be asked to the patients / proxies? The French version of the SWAL-QOL will be used

CONTACTS AND LOCATIONS:
Overall Officials: Yves Vandermeeren, MD, PhD, Principal Investigator — University Hospital of Mont-Godinne
Locations (1):
- University Hospital of Mont-Godinne : CHU Mont-Godinne UCL, Yvoir, Namur, Belgium